CLINICAL TRIAL: NCT06596655
Title: Implementation of Low-Cost Single-Use Flexible Bronchoscopes for Routine Interventional Pulmonary Procedures: A Feasibility Study
Brief Title: Single Use Bronchoscopes for Interventional Pulmonology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief, Section of Interventional Pulmonology, Division of Thoracic Surgery and Interventional Pulmonology,, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024P000471
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Bronchoscopic Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of single use bronchoscope (Experimental)
  Interventions: Device: Single use bronchoscope

INTERVENTIONS:
Device: Single use bronchoscope — Use of single use bronchoscopes for interventional pulmonology procedures instead of reusable bronchoscopes.

SUMMARY:
The goal of this pilot single-arm crossover trial is to investigate the feasibility and safety of using single-use flexible bronchoscopes (SUFB) for routine diagnostic and therapeutic interventional pulmonary procedures instead of reusable flexible bronchoscopes (RFB). The main questions it aims to answer are:

Was a decision to crossover from SUFB to RFB (at the discretion of the clinical bronchoscopist) made ?

Bronchoscopist's assessment of the SUFB for each procedure (using a Likert scale 0-10) including:

1. Overall assessment
2. Scope quality
3. Scope handling
4. Scope maneuverability
5. Tool compatibility
6. Suction
7. Lavage
8. Safety
9. Image quality

Participants will undergo bronchoscopy with single use bronchoscopes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to provide informed consent.

Exclusion Criteria:

1. Emergent procedure
2. Pregnancy
3. Study subjects have any diseases or conditions that interferes with safe completion of the biopsy including: cardiopulmonary instability; sensitivity to drugs that could be administered during bronchoscopy; active anticoagulation or antiplatelet therapy (warfarin, direct Xa inhibitors, thrombin inhibitors, low molecular weight heparin, unfractioned heparin, clopidogrel) not held adequately prior to the procedure; uncontrolled blood dyscrasias; concurrent pneumothorax or bullae.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of crossover from SUFB to RFB (at the discretion of the clinical bronchoscopist) | During the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No